CLINICAL TRIAL: NCT00959036
Title: A Seamless, Phase 1/2, Multiple Ascending Dose, Proof Of Concept Study Of ATN-103 Administered To Subjects With Active Rheumatoid Arthritis On A Background Of Methotrexate
Brief Title: Study Evaluating Multiple Doses Of ATN-103 In Subjects With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ablynx, a Sanofi company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3242K1-2000; B2271003
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Active Rheumatoid Arthritis
MeSH Terms: interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Treatment Group 1 (Experimental): ATN-103 10 mg every 4 weeks until week 12
  Interventions: Drug: ATN-103; Drug: Methotrexate
- Treatment Group 2 (Experimental): ATN-103 10 mg every 8 weeks until week 12
  Interventions: Drug: ATN-103; Drug: Methotrexate
- Treatment Group 3 (Experimental): ATN-103 30 mg every 4 weeks until week 12
  Interventions: Drug: ATN-103; Drug: Methotrexate
- Treatment Group 4 (Experimental): ATN-103 80 mg every 4 weeks until week 12
  Interventions: Drug: ATN-103; Drug: Methotrexate
- Treatment Group 5 (Experimental): ATN-103 80 mg every 8 weeks until week 12
  Interventions: Drug: ATN-103; Drug: Methotrexate
- Treatment Group 6 (Placebo Comparator): Placebo every 4 weeks
  Interventions: Drug: Placebo; Drug: Methotrexate

INTERVENTIONS:
Drug: ATN-103 — 10 mg every 4 weeks until week 12
  Arms: Treatment Group 1
Drug: ATN-103 — 10 mg every 8 weeks until week 12
  Arms: Treatment Group 2
Drug: ATN-103 — 30 mg every 4 weeks until week 12
  Arms: Treatment Group 3
Drug: ATN-103 — 80 mg every 4 weeks until week 12
  Arms: Treatment Group 4
Drug: ATN-103 — 80 mg every 8 weeks until week 12
  Arms: Treatment Group 5
Drug: Placebo — Placebo every 4 weeks
  Arms: Treatment Group 6
Drug: Methotrexate

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ATN-103 when administered to subjects with active rheumatoid arthritis compared with placebo. All subjects must be on a stable dose and route of methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of active rheumatoid arthritis on a stable background of methotrexate (7.5-25 mg weekly).

Exclusion Criteria:

* Any significant health problem other than rheumatoid arthritis
* Any clinically significant laboratory abnormalities
* Any prior use of B cell-depleting therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2009-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
American College of Rheumatology (ACR) 20 response at week 16 | 6 months

SECONDARY OUTCOMES:
Additional efficacy endpoints as measured by the number of swollen and tender joints, physician and patient global assessments of disease activity, ACR responses, DAS28, EULAR, and Health Outcome Assessments | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Josefin-Beate Holz, MD, Study Director — Ablynx, a Sanofi company
Locations (61):
- United States (35):
  - Investigational Site, Birmingham, Alabama
  - Investigational Site, Huntsville, Alabama
  - Investigational Site, Peoria, Arizona
  - Investigational Site, Scottsdale, Arizona
  - Investigational Site, Riverside, California
  - Investigational Site, Upland, California
  - Investigational Site, Bridgeport, Connecticut
  - Investigational Site, Newark, Delaware
  - Investigational Site, Lake Mary, Florida
  - Investigational Site, Ocala, Florida
  - Investigational Site, Orlando, Florida
  - Investigational Site, Port Orange, Florida
  - Investigational Site, Vero Beach, Florida
  - Investigational Site, Coeur d'Alene, Idaho
  - Investigational Site, Frederick, Maryland
  - Investigational Site, West Yarmouth, Massachusetts
  - Investigational Site, Lansing, Michigan
  - Investigational Site, Freehold, New Jersey
  - Investigational Site, Albuquerque, New Mexico
  - Investigational Site, Mineola, New York
  - Investigational Site, Charlotte, North Carolina
  - Investigational Site, Hickory, North Carolina
  - Investigational Site, Winston-Salem, North Carolina
  - Investigational Site, Columbus, Ohio
  - Investigational Site, Oklahoma City, Oklahoma
  - Investigational Site, Tulsa, Oklahoma
  - Investigational Site, Lake Oswego, Oregon
  - Investigational Site, Allentown, Pennsylvania
  - Investigational Site, Columbia, South Carolina
  - Investigational Site, Myrtle Beach, South Carolina
  - Investigational Site, Nashville, Tennessee
  - Investigational Site, Dallas, Texas
  - Investigational Site, Houston, Texas
  - Investigational Site, San Antonio, Texas
  - Investigational Site, Tacoma, Washington
- Belgium (2):
  - Investigational Site, Brussels, Belgium
  - Investigational Site, Leuven
- Canada (6):
  - Investigational Site, Winnipeg, Manitoba
  - Investigational Site, Kitchener, Ontario
  - Investigational Site, Ottawa, Ontario
  - Investigational Site, St. Catharines, Ontario
  - Investigational Site, Toronto, Ontario
  - Investigational Site, Québec, Quebec
- Investigational Site, Vogelsang, Gommern, Germany
- Hungary (2):
  - Investigational Site, Budapest
  - Investigational Site, Debrecen
- Russia (8):
  - Investigational Site, Kemerovo
  - Investigational Site, Moscow
  - Investigational Site, Novosibirsk
  - Investigational Site, Orenburg
  - Investigational Site, Petrozavodsk
  - Investigational Site, Ryazan
  - Investigational Site, Vladimir
  - Investigational Site, Yaroslavl
- Serbia (2):
  - Investigational Site, Belgrade, Serbia
  - Investigational Site, Niška Banja
- South Africa (3):
  - Investigational Site, Berea, KwaZulu-Natal
  - Investigational Site, Cape Town
  - Investigational Site, Pretoria
- Switzerland (2):
  - Investigational Site, Zurich, Canton of Zurich
  - Investigational Site, Chur